CLINICAL TRIAL: NCT06880263
Title: Using 360-Degree Immersive Virtual Reality to Enhance Nurses' Delirium Management Skills - A Randomized Controlled Trial
Brief Title: VR Training for Nurses' Delirium Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wen-Chii Tzeng, Professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B202505018
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: ICU Nurses, Delirium, Virtual Reality
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental)
  Interventions: Device: use 360 degree VR training
- Video group (Other)
  Interventions: Device: use 360 degree VR training

INTERVENTIONS:
Device: use 360 degree VR training — Participants will use Virtual Reality (VR) training

SUMMARY:
Background:

Delirium is an acute mental status change characterized by confusion, fluctuating symptoms, and inattention. It affects 11%-40% of hospitalized elderly patients and over 80% of mechanically ventilated ICU patients. Early detection and intervention are crucial in preventing adverse outcomes. The Confusion Assessment Method for the ICU (CAM-ICU) has been widely adopted in Taiwan for delirium screening. However, nurses' knowledge and skills in delirium assessment remain insufficient.

Objective:

This study aims to evaluate the effectiveness of a spherical video-based virtual reality (SVVR) training system in improving nurses' delirium assessment and management skills.

Methods:

A parallel-group randomized controlled trial will be conducted. Participants (nurses aged 20-65) will be recruited via social media and screened for eligibility. They will be randomly assigned to:

Intervention group: SVVR-based delirium training using a head-mounted display. Control group: Standard video-based training via YouTube. Pre- and post-intervention assessments will measure delirium knowledge, attitudes, assessment skills, learning motivation, and technology acceptance. Quantitative data will be analyzed using SPSS (Version 25) with t-tests, ANOVA, and chi-square tests. Qualitative data will be analyzed using thematic analysis.

Expected Outcome:

This study will determine whether immersive VR training enhances nurses' delirium management skills more effectively than conventional video training.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 65 years.
* Currently a licensed nurse and practicing.
* Willing to participate in this study and comply with the related procedures.
* Completed and signed the written informed consent form.

Exclusion Criteria:

* Nurse managers or nurses who do not directly care for patients, or nurses working in outpatient or community settings.
* Individuals with epilepsy, heart disease, or dizziness.
* Individuals with anxiety, panic disorder, or claustrophobia.
* Individuals with myopia greater than 600 degrees or those who have previously undergone eye surgery.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Chinese Version of Nurse's Assessment Ability Questionnaire in Delirium Subtypes | 20 mins
  VR group will get high score in assessment ability of Delirium Subtypes

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
If other relevant researchers need it, we will consider sharing the relevant information.